CLINICAL TRIAL: NCT00062335
Title: A Phase I Study On The Feasibility Of High Dose Three Dimensional Conformal Radiotherapy In Patients With Inoperable And Locally Advanced Non Small Cell Lung Cancer
Brief Title: High-Dose 3-Dimensional Conformal Radiation Therapy in Treating Patients With Inoperable Stage I, Stage II, or Stage IIIA Non-Small Cell Lung Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: low accrual
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: EORTC-22994; EORTC-22994
Record Dates: First submitted 2003-06-05; First posted 2003-06-06 (Estimated); Last update posted 2012-09-24 (Estimated); Status verified 2012-09

CONDITIONS: Lung Cancer
Keywords: stage I non-small cell lung cancer; stage II non-small cell lung cancer; stage IIIA non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Radiotherapy

INTERVENTIONS:
Radiation: radiation therapy

SUMMARY:
RATIONALE: Using computer systems that create a 3-dimensional picture of the tumor to plan treatment may enable doctors to provide more effective radiation therapy that will cause less damage to normal tissue.

PURPOSE: This phase I trial is studying the side effects and best dose of high-dose 3-dimensional conformal radiation therapy in treating patients with inoperable stage I, stage II, or stage IIIA non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the optimal dose of high-dose 3-dimensional conformal radiotherapy in patients with inoperable stage I, II, or IIIA non-small cell lung cancer who are treated according to the total lung volume irradiated.
* Determine the feasibility of this regimen, in terms of local control rates and incidence of distant metastases, in these patients.

OUTLINE: This is an open-label, nonrandomized, dose-escalation, multicenter study. Patients are assigned to 1 of 3 strata according to the total lung volume irradiated (less than 25% vs 25-37% vs over 37%).

* Stratum I: Patients undergo high-dose 3-dimensional (3-D) conformal radiotherapy 5 days a week for 6 weeks.
* Stratum II: Patients undergo high-dose 3-D conformal radiotherapy 5 days a week for 5.5-7 weeks.
* Stratum III: Patients undergo high-dose 3-D conformal radiotherapy 5 days a week for 5.5-6.5 weeks.

Cohorts of 6-15 patients in each stratum receive escalating dose intensities of high-dose 3-D conformal radiotherapy (either by increasing the total dose or by shortening treatment time) until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose at which 2 of 6, 2 of 15, or 3 of 30 patients experience dose-limiting toxicity.

Patients are followed at 1 month, at least every 2 months for 1 year, every 3 months for 1 year, and then every 6 months thereafter.

PROJECTED ACCRUAL: A total of 54-135 patients (18-45 per stratum) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed non-small cell lung cancer

  * Medically inoperable stage I or II disease
  * Stage III disease eligible provided the following are true:

    * No supraclavicular node involvement
    * No peripherally located lower lobe tumor AND contralateral upper mediastinal node involvement
* No distant metastasis
* No malignant pleural or pericardial effusion

PATIENT CHARACTERISTICS:

Age

* Not specified

Performance status

* WHO 0-2

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Not specified

Cardiovascular

* No prior myocardial infarction
* No prior complete bundle branch block
* No other prior cardiovascular disease resulting in New York Heart Association class III or IV heart disease
* No clinically significant cardiac arrhythmias
* No congestive heart failure

Pulmonary

* FEV_1 at least 1.2 L OR
* DLCO at least 60%

Other

* No other prior or concurrent malignancy except cured basal cell skin cancer or carcinoma in situ of the cervix
* No intractable or uncontrolled infection
* No psychological, familial, social, or geographical condition that would preclude study compliance and follow-up
* Able to tolerate a course of radiotherapy

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* At least 3 weeks since prior chemotherapy
* No prior anthracyclines
* No concurrent chemotherapy

Endocrine therapy

* Not specified

Radiotherapy

* No prior radiotherapy to the chest area

Surgery

* No prior therapeutic surgery to the chest area

Other

* No other prior therapy to the chest area

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2003-04; Primary Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose as measured by NCI-CTC v2.0 during treatment and up to 6 months after completion of radiotherapy

SECONDARY OUTCOMES:
Late toxicity measured every 2 months in year 1, then every 3 months in year 2, and then every 6 months thereafter
Disease progression measured every 2 months in year 1, then every 3 months in year 2, and then every 6 months thereafter

CONTACTS AND LOCATIONS:
Overall Officials: Jacques Bernier, MD, PhD, Study Chair — Istituto Oncologico della Svizzera Italiana - Ospedale San Giovanni
Locations (7):
- Belgium (3):
  - Institut Jules Bordet, Brussels
  - Academisch Ziekenhuis der Vrije Universiteit Brussel, Brussels
  - Akademisch Ziekenhuis Gent, Ghent
- France (3):
  - Centre Regional de Lutte Contre le Cancer - Centre Val d'Aurelle, Montpellier
  - Centre Antoine Lacassagne, Nice
  - Institut Curie - Section Medicale, Paris
- Centre Hospitalier Universitaire Vaudois, Lausanne, Switzerland